CLINICAL TRIAL: NCT00003174
Title: Phase I Clinical Evaluation of Bryostatin 1 in Combination With 2-CdA in Patients With Relapsed CLL
Brief Title: Bryostatin 1 Plus Cladribine in Treating Patients With Relapsed Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065984; P30CA022453 (NIH); WSU-C-1388; NCI-T97-0016
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Leukemia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — bryostatin 1; Cladribine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bryostatin 1
Drug: cladribine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of cladribine when given with bryostatin 1 in treating patients with relapsed chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of cladribine when administered after bryostatin 1 in patients with relapsed chronic lymphocytic leukemia.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of cladribine.

Patients receive bryostatin 1 IV continuously on days 1-3 immediately followed by cladribine IV continuously on days 4-8. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Patients who achieve complete remission (CR) receive 2 additional courses past CR.

Cohorts of 3-6 patients receive escalating dose levels of cladribine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 3 weeks.

PROJECTED ACCRUAL: A minimum of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of relapsed chronic lymphocytic leukemia

  * Intermediate- or high-risk (stage I-IV) disease
* Intermediate-risk patients must have active disease, defined by at least 1 of the following criteria:

  * Presence of any 1 of the following disease-related B symptoms:

    * 10% or more loss of body weight within the past 6 months
    * Extreme fatigue
    * Fever greater than 100 degrees Fahrenheit without evidence of infection
    * Night sweats
  * Massive (greater than 6 cm below left costal margin) or progressive splenomegaly
  * Massive (greater than 10 cm in longest diameter) or progressive lymphadenopathy
  * Progressive lymphocytosis with an increase of more than 50% over a 2-month period or anticipated doubling time of less than 12 months
  * Progressive bone marrow failure as manifested by the development or worsening of anemia and/or thrombocytopenia
  * Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroids
* Failed 1-2 prior front-line regimens
* Failed prior fludarabine
* Ineligible for any known treatment of higher potential efficacy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* See Disease Characteristics
* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* Transaminases less than 2.5 times normal

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No history of severe coronary artery disease, cardiomyopathy, uncontrolled congestive heart failure, or arrhythmias

Neurologic:

* No prior drug-related neurotoxicity
* No other neurologic disorder

Other:

* Not pregnant or nursing
* Fertile patients must use effective barrier or non-hormonal contraception during and for 2 months after study participation
* No HIV infection
* No AIDS

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow transplantation

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (8 weeks for mitomycin or nitrosoureas) and recovered

Endocrine therapy:

* See Disease Characteristics
* No concurrent steroids
* No concurrent hormonal contraceptives

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No other concurrent therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 1998-05; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayad M. Al-Katib, MD, FACP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (3):
- United States (3):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan

REFERENCES:
- [Background] Ahmad I, Al-Katib AM, Beck FW, Mohammad RM. Sequential treatment of a resistant chronic lymphocytic leukemia patient with bryostatin 1 followed by 2-chlorodeoxyadenosine: case report. Clin Cancer Res. 2000 Apr;6(4):1328-32. PMID 10778958